CLINICAL TRIAL: NCT06752252
Title: Ultrasound Guided Paravertebral Block Versus Erector Spinae Plane Block for Postoperative Analgesia After Inguinal Hernia Repair in Pediatric Patients: a Randomized Clinical Trial
Brief Title: Ultrasound Guided Paravertebral Block Versus Erector Spinae Block for Postoperative Analgesia After Inguinal Hernia Repair in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 866
Record Dates: First submitted 2024-12-21; First posted 2024-12-30 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Analgesia, Postoperative
Keywords: postoperative analgesia; ultrasound guided paravertebral block; ultrasound guided erector spinae plane block; inguinal hernia repair in pediatric
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Postoperative analgesia after inguinal hernia repair in pediatric by ultrasound guided paravertebral block or erector spinae block
Who Masked: Participant, Outcomes Assessor
Masking Description: anesthetist not sharing in the study will assess patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group paravertebral (PVB) block (Active Comparator): In the lateral decubitus and after sterilization and identifying the level of T10 ,linear ultrasound probe will be placed in the midline over the spinous process at the chosen level, then the probe will be moved laterally to view the lamina and hyperechoic transverse process ,the pleural should be visible as a bright white line .The needle should be inserted in -plane from lateral to medial and the needle tip should end in a hypoechoic triangular space .Correct needle placement should be confirmed by anterior displacement of pleura with injection of small volume of saline then 0.5 ml/kg of a mixture of 0.25 ℅ bupivacaine and 1℅ lidocaine (1:1) will be injected
  Interventions: Procedure: ultrasound guided paravertebral block
- Group erector spinae plane (ESP) block (Active Comparator): In the lateral decubitus position ,after sterilization, the linear ultrasound probe will be placed over transverse process of T10 ,after optimizing the image in sagittal or transverse scanning ,A 50 mm 22-G needle will be placed under the erector spinae muscle in -in plane orientation until it contacted T8 transverse process in the cranial caudal direction ,after hydro dissection and confirmation that the tip of the needle is between the transverse process and the fascia of the erector spinae muscle group, 0.5 ml/kg of a mixture of 0.25 ℅bupivacaine and 1℅ lidocaine (1:1) will be injected and the surgery will be started after 15 min
  Interventions: Procedure: Ultrasound guided erector spinae plane block
- Control group (group C) (Active Comparator): will receive standard general anesthesia with pain management protocol without regional block. Pain management protocol for all patients will include IV paracetamol 15 mg/kg every 6 hrs. (max dose for children <50 kg is 60 mg/kg daily and if body weight ≥ 50 kg max dose is 4 gm daily) . Ibuprofen will be given as rescue analgesia 10 mg/kg IV if MOPS was > 3 at rest or after movement and can be repeated every 6 hrs not exceeding 400 mg/dose and max daily dose 40 mg/kg.
  Interventions: Procedure: control group C

INTERVENTIONS:
Procedure: ultrasound guided paravertebral block — after sterilization and identifying the level of T10 ,linear ultrasound probe will be placed in the midline over the spinous process at the chosen level, then the probe will be moved laterally to view the lamina and hyperechoic transverse process ,the pleural should be visible as a bright white line .The needle should be inserted in -plane from lateral to medial and the needle tip should end in a hypoechoic triangular space. Correct needle placement should be confirmed by anterior displacement of pleura with injection of small volume of saline then 0.5 ml/kg of a mixture of 0.25 ℅ bupivacaine and 1℅ lidocaine (1:1) will be injected
  Arms: Group paravertebral (PVB) block
Procedure: Ultrasound guided erector spinae plane block — After sterilization, the linear ultrasound probe will be placed over transverse process of T10 ,after optimizing the image in sagittal or transverse scanning ,A 50 mm 22-G needle will be placed under the erector spinae muscle in -in plane orientation until it contacted T8 transverse process in the cranial caudal direction ,after hydro dissection and confirmation that the tip of the needle is between the transverse process and the fascia of the erector spinae muscle group, 0.5 ml/kg of a mixture of 0.25 ℅bupivacaine and 1℅ lidocaine (1:1) will be injected
  Arms: Group erector spinae plane (ESP) block
Procedure: control group C — will receive standard general anesthesia with pain management protocol without regional block.
  Arms: Control group (group C)

SUMMARY:
The aim of the study is to compare postoperative analgesia in pediatric patients undergoing inguinal hernia repair by comparing the efficacy of ultrasound guided paravertebral block versus ultrasound guided erector spinae plane block.

DETAILED DESCRIPTION:
* To assess the total amount of rescue analgesic consumption in the first 24 hours post-operatively in each group.
* To measure the time of first request of rescue analgesia and to assess pain intensity at rest (static) and after movement or coughing (dynamic) using 10 points Modified Objective Pain Score (MOPS).
* To record the incidence of complications (hematoma, local anesthetic toxicity, pneumothorax, infection, hypotension, epidural or intrathecal spread).
* Over all parent's satisfaction: The parents will be asked to rate the overall degree of satisfaction of the analgesia by using a 5-points likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia).

ELIGIBILITY:
Inclusion Criteria:

1 - Parents acceptance

2. Age: preschool and school age child (24 months-12 years old).

3. Sex: both sex (males or females).

4. Physical status: ASA 1& II.

5. Type of operation: elective unilateral inguinal hernia repair

Exclusion Criteria:

1- Patient with any contraindications of regional blocks (as coagulopathy or local infection at injection site)

2. Patients with known history of allergy to the study drugs (bupivacaine and lidocaine).

3. Advanced hepatic, renal, cardiovascular, neurologic and respiratory diseases.

Ages: 24 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 158 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The total amount of rescue analgesia (Ibuprofen consumption) | for 24 hours postoperative
  The total consumption of rescue analgesia (Ibuprofen consumption) postoperative

SECONDARY OUTCOMES:
Pain intensity at rest (static) and after movement or coughing (dynamic) | 0 minutes immediate postoperative ( on arrival to PACU), 30 minutes, 1hs, 2hs, 4hs, 8hs, 12 hrs and 24hs postoperatively
  by using 10 points Modified Objective Pain Score (MOPS)(0=no pain, 1-3=mild pain, 4-6=moderate pain, and 7-10= sever pain)
The time to first request of rescue analgesia (Ibuprofen) | for 24 hours postoperative
  the time from giving block till time of first request of ibuprofen when MOPS > 3 at rest or after movement
The total number of patients requiring additional dose of intraoperative fentanyl. | during operation period
  Number of patients receive additional dose of intra operative fentanyl ( increase in the mean blood pressure or heart rate 20% above base line readings, fentanyl in a dose 0.5 mcg/kg will be given to the patient)
To record the incidence of complications | 24 hours postoperative
  To record the incidence of complications (hematoma, local anesthetic toxicity, pneumothorax, infection, hypotension, epidural or intrathecal spread)
Over all parent's satisfaction | 24 hours postoperative
  The parents will be asked to rate the overall degree of satisfaction of the analgesia by using a 5-points likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - faculty of human medicine, Zagazig university hospitals, El Sharkia
  - Faculty of Human Medicine, Zagazig University, El Sharkia

IPD SHARING:
Plan to Share IPD: No